CLINICAL TRIAL: NCT05751954
Title: Influence of Weight-bearing Mechanical Axis on Foot and Ankle in Patients Following Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinic for Orthopedics Lovran (Other)
Responsible Party: Principal Investigator, Antea Buterin, MD, Clinic for Orthopedics Lovran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEH01
Record Dates: First submitted 2019-08-31; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Total Knee Artroplasty
Keywords: weight-bearing mechanical axis; total knee arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Label (Other): All patients who undergo total knee arthroplasty and met inclusion and exclusion criteria
  Interventions: Radiation: Postero-anterior weight-bearing full-leg radiograph; Device: Pedobarographic analysis

INTERVENTIONS:
Radiation: Postero-anterior weight-bearing full-leg radiograph — Full leg standing X ray of the involved lower extremity (postero-anterior direction)
Device: Pedobarographic analysis — Foot pressure analysis during gait on pedobarographic device

SUMMARY:
This comprehensive scientific research will investigate the influence of the weight-bearing mechanical axis on foot and ankle following total knee arthroplasty. Few studies have monitored the outcome of surgical treatment using similair methods, and consequently the aim of this study was to evaluate the change in upper and lower leg load by analyzing radiographic recordings and pedobarographic measurements after the implantation of total knee endoprosthesis. In addition to objective instruments, knee and foot questionnaires will be used to describe the functional outcome of the operation of the subjects. The practical contribution of this research lies in the prediction of possible changes in the joints of the feet depending on the type of knee deformity (varus / valgus). Our research will consist of: analysis of postero-anterior radiographs of the lower extremity (weight-bearing) preoperatively and at the follow-up three months postoperatively, pedobarographic analyzes preoperatively and at the control examination three months postoperatively, analysis of personal data (age, gender, weight and height, operated side) and completion of functional standardized questionnaires (AOFAS, KOOS) preoperatively, and at the screening three months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* knee varus or valgus deformity 5 degrees or more

Exclusion Criteria:

* previous surgery which included corrective osteotomies, osteosynthesis or arthrodesis of the knee, ankle and foot.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight-bearing mechanical axis | 1 year

SECONDARY OUTCOMES:
Pedobarographic analysis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Orthopeadics and Traumatology Lovran, Lovran, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided